CLINICAL TRIAL: NCT03759470
Title: Evaluation of Different Methods for Rapid Diagnosis of Meningitis in Assiut University Hospital
Brief Title: Evaluation of Different Methods for Diagnosis of ME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Doha Fahmy (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Doha Fahmy, Principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Doha Fahmy
Record Dates: First submitted 2018-11-20; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Diagnoses Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation of different methods for diagnosis of meningitis: The CSF samples will be stored at -80°C until testing . CSF specimens will be prepared for GS and culture examinations by centrifugation at 3,000 rpm for 10 minutes at room temperaturetemperature.Culture will be performed by inoculating 1-2 drops of CSF sediment directly onto each of the following agar plates: horse-blood agar, Thayer-Martin agar, choc- olate agar and Sabouraud agar. Moreover, a broth tube (brain-heart infusion, BHI) will be inoculated with one drop of the sediment. Agar plates and broth will be incubated for 1 to 5 days at 35-37°C (with ~5% CO2, or in a candle-jar, for Thayer-Martin and chocolate agar) .
  In addition to GS and culture method , India ink test and culture and latex agglutination test (LAT). LAT assay will be performed on CSF samples using Latex-antigen detection system kit..
  Interventions: Diagnostic Test: CSF examination

INTERVENTIONS:
Diagnostic Test: CSF examination — The CSF samples will be stored at -80°C until testing . CSF specimens will be prepared for GS and culture examinations by centrifugation at 3,000 rpm for 10 minutes at room temperature. Culture will be performed by inoculating 1-2 drops of CSF sediment directly onto each of the following agar plates: horse-blood agar, Thayer-Martin agar, choc- olate agar and Sabouraud agar. Moreover, a broth tube (brain-heart infusion, BHI) will be inoculated with one drop of the sediment. Agar plates and broth will be incubated for 1 to 5 days at 35-37°C (with ~5% CO2, or in a candle-jar, for Thayer-Martin and chocolate agar) .
  In addition to GS and culture method , India ink test and culture and latex agglutination test (LAT). LAT assay will be performed on CSF samples using Latex-antigen detection system kit.

SUMMARY:
Bacterial meningitis occurs in about 3 people per 100,000 annually in Western countries. .

DETAILED DESCRIPTION:
meningitis is a notifiable disease in many countries, the exact incidence rate is unknown. In 2013 meningitis resulted in 303,000 deaths - down from 464,000 deaths in 1990. In 2010 it was estimated that meningitis resulted in 420,000 deaths, excluding cryptococcal meningitis.

Bacterial meningitis occurs in about 3 people per 100,000 annually in Western countries. Population-wide studies have shown that viral meningitis is more common, at 10.9 per 100,000, and occurs more often in the summer. In Brazil, the rate of bacterial meningitis is higher, at 45.8 per 100,000 annually.Sub-Saharan Africa has been plagued by large epidemics of meningococcal meningitis for over a century,leading to it being labeled the "meningitis belt". Epidemics typically occur in the dry season (December to June), and an epidemic wave can last two to three years, dying out during the intervening rainy seasons.Attack rates of 100-800 cases per 100,000 are encountered in this area, which is poorly served by medical care. These cases are predominantly caused by meningococci.The largest epidemic ever recorded in history swept across the entire region in 1996-1997, causing over 250,000 cases and 25,000 deaths.

Meningococcal disease occurs in epidemics in areas where many people live together for the first time, such as army barracks during mobilization, college campuses and the annual Hajj pilgrimage. Although the pattern of epidemic cycles in Africa is not well understood, several factors have been associated with the development of epidemics in the meningitis belt. They include: medical conditions (immunological susceptibility of the population), demographic conditions (travel and large population displacements), socioeconomic conditions (overcrowding and poor living conditions), climatic conditions (drought and dust storms), and concurrent infections (acute respiratory infections).

There are significant differences in the local distribution of causes for bacterial meningitis. For instance, while N. meningitides groups B and C cause most disease episodes in Europe, group A is found in Asia and continues to predominate in Africa, where it causes most of the major epidemics in the meningitis belt, accounting for about 80% to 85% of documented meningococcal meningitis cases.

Infections that involve the central nervous system (CNS), such as meningitis/encephalitis (ME), are severe clinical conditions associated with high rates of morbidity and mortality as well as significant long-term sequelae . acute inflammation of the protective membranes covering the brain and spinal cord, known collectively as the meninges.The most common symptoms are fever, headache, and neck stiffness.Other symptoms include confusion or altered consciousness, vomiting, and an inability to tolerate light or loud noises. Young children often exhibit only nonspecific symptoms, such as irritability, drowsiness, or poor feeding.If a rash is present, it may indicate a particular cause of meningitis; for instance, meningitis caused by meningococcal bacteria may be accompanied by a characteristic rash. The inflammation may be caused by infection with viruses, bacteria, or other microorganisms, and less commonly by certain drugs.Meningitis can be life-threatening because of the inflammation's proximity to the brain and spinal cord; therefore, the condition is classified as a medical emergency. A lumbar puncture can diagnose or exclude meningitis.A needle is inserted into the spinal canal to collect a sample of cerebrospinal fluid (CSF), which envelops the brain and spinal cord. The CSF is examined in a medical laboratory.

Some forms of meningitis are preventable by immunization with the meningococcal, mumps, pneumococcal, and Hib vaccines.Giving antibiotics to people with significant exposure to certain types of meningitis may also be useful.The first treatment in acute meningitis consists of promptly giving antibiotics and sometimes antiviral drugs.Corticosteroids can also be used to prevent complications from excessive inflammation. Meningitis can lead to serious long-term consequences such as deafness, epilepsy, hydrocephalus, or cognitive deficits, especially if not treated quickly.

most common symptom of meningitis is a severe headache, occurring in almost 90% of cases of bacterial meningitis, followed by nuchal rigidity (the inability to flex the neck forward passively due to increased neck muscle tone and stiffness). The classic triad of diagnostic signs consists of nuchal rigidity, sudden high fever, and altered mental status; however, all three features are present in only 44-46% of bacterial meningitis cases.If none of the three signs are present, acute meningitis is extremely unlikely.Other signs commonly associated with meningitis include photophobia (intolerance to bright light) and phonophobia (intolerance to loud noises). Small children often do not exhibit the aforementioned symptoms, and may only be irritable and look unwell.The fontanelle (the soft spot on the top of a baby's head) can bulge in infants aged up to 6 months. Other features that distinguish meningitis from less severe illnesses in young children are leg pain, cold extremities, and an abnormal skin color.

Nuchal rigidity occurs in 70% of bacterial meningitis in adults. Other signs include the presence of positive Kernig's sign or Brudziński sign. Kernig's sign is assessed with the person lying supine, with the hip and knee flexed to 90 degrees. In a person with a positive Kernig's sign, pain limits passive extension of the knee. A positive Brudzinski's sign occurs when flexion of the neck causes involuntary flexion of the knee and hip. Although Kernig's sign and Brudzinski's sign are both commonly used to screen for meningitis, the sensitivity of these tests is limited.They do, however, have very good specificity for meningitis: the signs rarely occur in other diseases. Another test, known as the "jolt accentuation maneuver" helps determine whether meningitis is present in those reporting fever and headache. A person is asked to rapidly rotate the head horizontally; if this does not make the headache worse, meningitis is unlikely.

Other problems can produce symptoms similar to those above, but from non-meningitic causes. This is called meningism or pseudomeningitis.

Meningitis caused by the bacterium Neisseria meningitidis (known as "meningococcal meningitis") can be differentiated from meningitis with other causes by a rapidly spreading petechial rash, which may precede other symptoms.The rash consists of numerous small, irregular purple or red spots ("petechiae") on the trunk, lower extremities, mucous membranes, conjuctiva, and (occasionally) the palms of the hands or soles of the feet. The rash is typically non-blanching; the redness does not disappear when pressed with a finger or a glass tumbler. Although this rash is not necessarily present in meningococcal meningitis, it is relatively specific for the disease; it does, however, occasionally occur in meningitis due to other bacteria. Other clues on the cause of meningitis may be the skin signs of hand, foot and mouth disease and genital herpes, both of which are associated with various forms of viral meningitis.

Additional problems may occur in the early stage of the illness. These may require specific treatment, and sometimes indicate severe illness or worse prognosis. The infection may trigger sepsis, a systemic inflammatory response syndrome of falling blood pressure, fast heart rate, high or abnormally low temperature, and rapid breathing. Very low blood pressure may occur at an early stage, especially but not exclusively in meningococcal meningitis; this may lead to insufficient blood supply to other organs.Disseminated intravascular coagulation, the excessive activation of blood clotting, may obstruct blood flow to organs and paradoxically increase the bleeding risk. Gangrene of limbs can occur in meningococcal disease.Severe meningococcal and pneumococcal infections may result in hemorrhaging of the adrenal glands, leading to Waterhouse-Friderichsen syndrome, which is often fatal.

The brain tissue may swell, pressure inside the skull may increase and the swollen brain may herniate through the skull base. This may be noticed by a decreasing level of consciousness, loss of the pupillary light reflex, and abnormal posturing.The inflammation of the brain tissue may also obstruct the normal flow of CSF around the brain (hydrocephalus).Seizures may occur for various reasons; in children, seizures are common in the early stages of meningitis (in 30% of cases) and do not necessarily indicate an underlying cause.Seizures may result from increased pressure and from areas of inflammation in the brain tissue. Focal seizures (seizures that involve one limb or part of the body), persistent seizures, late-onset seizures and those that are difficult to control with medication indicate a poorer long-term outcome.

Inflammation of the meninges may lead to abnormalities of the cranial nerves, a group of nerves arising from the brain stem that supply the head and neck area and which control, among other functions, eye movement, facial muscles, and hearing. Visual symptoms and hearing loss may persist after an episode of meningitis.Inflammation of the brain (encephalitis) or its blood vessels (cerebral vasculitis), as well as the formation of blood clots in the veins (cerebral venous thrombosis), may all lead to weakness, loss of sensation, or abnormal movement or function of the part of the body supplied by the affected area of the brain.

Meningitis is typically caused by an infection with microorganisms. Most infections are due to viruses,with bacteria, fungi, and protozoa being the next most common causes. It may also result from various non-infectious causes. The term aseptic meningitis refers to cases of meningitis in which no bacterial infection can be demonstrated. This type of meningitis is usually caused by viruses but it may be due to bacterial infection that has already been partially treated, when bacteria disappear from the meninges, or pathogens infect a space adjacent to the meninges (e.g. sinusitis). Endocarditis (an infection of the heart valves which spreads small clusters of bacteria through the bloodstream) may cause aseptic meningitis. Aseptic meningitis may also result from infection with spirochetes, a group of bacteria that includes Treponema pallidum (the cause of syphilis) and Borrelia burgdorferi (known for causing Lyme disease). Meningitis may be encountered in cerebral malaria (malaria infecting the brain) or amoebic meningitis, meningitis due to infection with amoebae such as Naegleria fowleri, contracted from freshwater sources.

In premature babies and newborns up to three months old, common causes are group B streptococci (subtypes III which normally inhabit the vagina and are mainly a cause during the first week of life) and bacteria that normally inhabit the digestive tract such as Escherichia coli (carrying the K1 antigen). Listeria monocytogenes (serotype IVb) is transmitted by the mother before birth and may cause meningitis in the newborn.

Older children are more commonly affected by Neisseria meningitidis (meningococcus) and Streptococcus pneumoniae (serotypes 6, 9, 14, 18 and 23) and those under five by Haemophilus influenzae type B (in countries that do not offer vaccination).

Tuberculous meningitis, which is meningitis caused by Mycobacterium tuberculosis, is more common in people from countries in which tuberculosis is endemic, but is also encountered in persons with immune problems, such as AIDS.

Recurrent bacterial meningitis may be caused by persisting anatomical defects, either congenital or acquired, or by disorders of the immune system.Anatomical defects allow continuity between the external environment and the nervous system. The most common cause of recurrent meningitis is a skull fracture, particularly fractures that affect the base of the skull or extend towards the sinuses and petrous pyramids. Approximately 59% of recurrent meningitis cases are due to such anatomical abnormalities, 36% are due to immune deficiencies (such as complement deficiency, which predisposes especially to recurrent meningococcal meningitis), and 5% are due to ongoing infections in areas adjacent to the meninges.

Viruses that cause meningitis include enteroviruses, herpes simplex virus (generally type 2, which produces most genital sores; less commonly type 1), varicella zoster virus (known for causing chickenpox and shingles), mumps virus, HIV, and LCMV.[20] Mollaret's meningitis is a chronic recurrent form of herpes meningitis; it is thought to be caused by herpes simplex virus type 2.

There are a number of risk factors for fungal meningitis, including the use of immunosuppressants (such as after organ transplantation), HIV/AIDS, and the loss of immunity associated with aging.It is uncommon in those with a normal immune system but has occurred with medication contamination.Symptom onset is typically more gradual, with headaches and fever being present for at least a couple of weeks before diagnosis.The most common fungal meningitis is cryptococcal meningitis due to Cryptococcus neoformans. In Africa, cryptococcal meningitis is now the most common cause of meningitis in multiple studies,and it accounts for 20-25% of AIDS-related deaths in Africa.Other less common fungal pathogens which can cause meningitis include: Coccidioides immitis, Histoplasma capsulatum, Blastomyces dermatitidis, and Candida species.

A parasitic cause is often assumed when there is a predominance of eosinophils (a type of white blood cell) in the CSF. The most common parasites implicated are Angiostrongylus cantonensis, Gnathostoma spinigerum, Schistosoma, as well as the conditions cysticercosis, toxocariasis, baylisascariasis, paragonimiasis, and a number of rarer infections and noninfective conditions.

Untreated, bacterial meningitis is almost always fatal. Viral meningitis, in contrast, tends to resolve spontaneously and is rarely fatal. With treatment, mortality (risk of death) from bacterial meningitis depends on the age of the person and the underlying cause. Of newborns, 20-30% may die from an episode of bacterial meningitis. This risk is much lower in older children, whose mortality is about 2%, but rises again to about 19-37% in adults.Risk of death is predicted by various factors apart from age, such as the pathogen and the time it takes for the pathogen to be cleared from the cerebrospinal fluid,the severity of the generalized illness, a decreased level of consciousness or an abnormally low count of white blood cells in the CSF. Meningitis caused by H. influenzae and meningococci has a better prognosis than cases caused by group B streptococci, coliforms and S. pneumonia. In adults, too, meningococcal meningitis has a lower mortality (3-7%) than pneumococcal disease.

In children there are several potential disabilities which may result from damage to the nervous system, including sensorineural hearing loss, epilepsy, learning and behavioral difficulties, as well as decreased intelligence. These occur in about 15% of survivors.Some of the hearing loss may be reversible. In adults, 66% of all cases emerge without disability. The main problems are deafness (in 14%) and cognitive impairment (in 10%).

Tuberculous meningitis in children continues to be associated with a significant risk of death even with treatment (19%), and a significant proportion of the surviving children have ongoing neurological problems. Just over a third of all cases survives with no problems.

ELIGIBILITY:
Inclusion Criteria:

* childrens admitted inside Assiut university hospital with ME and fullfilling it's symptoms and signs.

Exclusion Criteria:

* -Childrens with symptoms and signs that are not consistenet with ME.

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Childrens with signs and symptoms of meningitis admitted in assiut university hospital in 2019
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of CSF and blood samples in diagnosis of meningitis in children's. | One year
  The CSF samples will be stored at -80°C until testing . CSF specimens will be prepared for GS and culture examinations by centrifugation at 3,000 rpm for 10 minutes at room temperature. When dry, the smear will be fixed stained and finally observed by light microscopy with a 100X objective. Culture will be performed by inoculating 1-2 drops of CSF sediment directly onto each of the following agar plates: horse-blood agar, Thayer-Martin agar, choc- olate agar and Sabouraud agar. Moreover, a broth tube (brain-heart infusion, BHI) will be inoculated with one drop of the sediment. Agar plates and broth will be incubated for 1 to 5 days at 35-37°C (with ~5% CO2, or in a candle-jar, for Thayer-Martin and chocolate agar) .
  In addition to GS and culture method , India ink test and culture and latex agglutination test (LAT). LAT assay will be performed on CSF samples using Latex-antigen detection system kit.